CLINICAL TRIAL: NCT06091748
Title: An Open-label, Single Arm Clinical Trial of Gallium (68Ga) Edotreotide PET-CT Scan for Imaging Patients With Gastrointestinal Pancreatic Neuroendocrine Tumors
Brief Title: Gallium (68Ga) Edotreotide PET/CT for Imaging Patients With Gastrointestinal Pancreatic Neuroendocrine Tumors
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HRFS-Q-2010-301
Record Dates: First submitted 2023-10-16; First posted 2023-10-19 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Advanced Gastroenteropancreatic Neuroendocrine Tumor
MeSH Terms: interventions — Ga(III)-DOTATOC

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PET/CT imaging with 68Ga-DOTATOC (Experimental)
  Interventions: Drug: 68Ga-DOTATOC

INTERVENTIONS:
Drug: 68Ga-DOTATOC — Detection of somatostatin positive lesions in GEP-NETs

SUMMARY:
This is a single-arm imaging study using DOTATOC peptide, labelled with the Gallium (68Ga) tracer.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent;
2. 18~75 years old,male or female；
3. ECOG performance status 0 or 1;
4. Confirmed or suspicion of GEP-NET.

Exclusion Criteria:

1. Unable to lie flat for the entire imaging duration (e.g. persistent cough, claustrophobia, severe arthritis, etc.), unable to enter the PET/CT device;
2. Individuals planning to be pregnant, and lactating women;
3. Individuals with concurrent active infections or with unexplained fever >38.5°C for more than 1 hour during the screening period or prior to administration of investigational medication.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-02-22 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of 68Ga-DOTATOC PET-CT Imaging for Detection of Somatostatin Receptor Positive GEP-NET | 12 months
  The number of patients with SSTR (+) GEP-NETs disease that was confirmed by imaging using 68Ga-DOTATOC PET/CT and Standard of Truth
Specificity of 68Ga-DOTATOC PET-CT Imaging for Detection of Somatostatin Receptor Positive GEP-NET | 12 months
  The number of patients who have no SSTR (+) GEP-NETs disease that was confirmed by imaging using 68Ga-DOTATOC PET/CT and Standard of Truth

SECONDARY OUTCOMES:
Incidence and severity of AE and SAE | up to 1 year follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided